CLINICAL TRIAL: NCT06795204
Title: A Randomized, Positive and Placebo-Controlled Study to Evaluate the Effects of HSK3486 Administration on Cardiac Repolarization in Healthy Subjects
Brief Title: Effects of HSK3486 on Cardiac Repolarization in Health Subjects (TQT)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Haisco-USA Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSK3486-112; NCT06379867 (obsolete NCT alias)
Record Dates: First submitted 2025-01-22; First posted 2025-01-27 (Actual); Results first posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Anesthesia; Adverse Effect; Cardiac Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — HSK3486; Moxifloxacin

STUDY DESIGN:
Intervention Model Description: Randomized, blinded (except moxifloxacin hydrochloride tablet), placebo and positive-controlled, 6-sequence, three-period crossover design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- HSK3486( study drug) (Experimental): One time, 0.4 mg/kg, IV bolus administration for 30 (±5) seconds
  Interventions: Drug: HSK3486
- Placebo (Placebo Comparator): One time, IV bolus administration for 30 (±5) seconds
  Interventions: Drug: Placebo
- Moxifloxacin hydrochloride (Active Comparator): One time, 0.4 g oral administration with 240 mL of warm water on an empty stomach.
  Interventions: Drug: Moxifloxacin Hydrochloride

INTERVENTIONS:
Drug: HSK3486 — Study Drug
  Other Names: Cipepofol
  Arms: HSK3486( study drug)
Drug: Moxifloxacin Hydrochloride — Positive Control
  Arms: Moxifloxacin hydrochloride
Drug: Placebo — Negative Control
  Arms: Placebo

SUMMARY:
To assess the effects of a single IV bolus of HSK3486 single dose on cardiac repolarization (QTc interval of the electrocardiogram, and to evaluate the safety and tolerability of a single IV bolus of HSK3486 in healthy subjects

DETAILED DESCRIPTION:
This is a single-center, randomized, blinded (except moxifloxacin hydrochloride tablet), placebo and positive controlled study with a 6-sequence, three-period crossover design in healthy subjects. A blinded design is used for administration of HSK3486 and placebo, and an open-label design is used for moxifloxacin hydrochloride tablet.

Subjects meet the including criteria and none of exclusion criteria are randomized in equal proportion to one of 6 dosing sequences (see Table 2 for dosing sequences), and the study procedure consisted of 3 periods, with washout period of 5 days between periods.

Subjects are closely monitored on vital sign checking, 12-lead ECG, and Holter collection through out each treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and comply with protocol requirements and was voluntarily sign written informed consent form (ICF).
2. Healthy participants at age from 18 to 45 years old (inclusive) at Screening.
3. Male body weight ≥50 kg, female body weight ≥45 kg, with a body mass index BMI of 19~28 kg/m2 (inclusive).
4. Left Ventricular Ejection Fraction (LVEF)≥50%.

Exclusion Criteria:

1. Past or present clinically significant systemic disease as judged by the Investigator including, but not limited to psychiatric, neurologic, pulmonary, respiratory, cardiac, gastrointestinal, genitourinary, renal, hepatic, metabolic, endocrinologic, hematological, or autoimmune disorders.
2. History of allergy to egg or egg products, soybean or soy products.
3. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance. History of allergy to HSK3486 or moxifloxacin or its investigational product excipients, or history of specific allergies (asthma, urticaria, eczema, etc.), or history of tendinitis or tendon rupture due to moxifloxacin or any other quinolone drug.
4. Clinically significant infection/injury/disease within 1 month prior to dosing.
5. Current or recent (< 6 months from screening) hepatobiliary disease.
6. Current or history of seizure disorder, including alcohol- or stimulant-related seizure, febrile seizure, or significant family history of idiopathic seizure disorder.
7. Family history of sudden death at <50 years of age.
8. History of unexplained loss of consciousness, unexplained syncope, unexplained irregular heartbeats or palpitations, clinically significant head injury.
9. Pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, or conditions that could interfere with the absorption, metabolism, and/or excretion of study drug (e.g., history of bariatric surgery or intestinal bypass surgery; simple uncomplicated appendectomies and hernia repairs are allowed, but cholecystectomy is not allowed).
10. Positive test results for hepatitis B surface antigen, hepatitis C antibody, treponema pallidum antibody, human immunodeficiency virus (HIV) antigen/antibody combination test.
11. Subjects with previous or suspected difficult airway (e.g., modified Mallampati score III- IV, congenital microglossia, mandibular dysplasia), or respiratory insufficiency, history of obstructive pulmonary disease, history of asthma, sleep apnea syndrome; history of failed tracheal intubation; history of bronchospasm requiring treatment within 3 months prior to screening; acute respiratory infection, and with obvious symptoms such as fever, wheezing, nasal congestion or cough within 1 week prior to baseline.
12. Knowledge of any kind of cardiovascular disorder/condition/procedure known to increase the possibility of QT prolongation or history of risk factors for torsade de pointes (e.g., heart failure, hypokalemia, hypomagnesemia, congenital Long QT syndrome, or family history of Long QT Syndrome).
13. Laboratory tests at screening or baseline judged clinically significant by the investigator, including, but not limited to, alanine aminotransferase (ALT) or aspartate aminotransferase or aspartate aminotransferase (AST) > 1.2 × upper limit of normal (ULN)(the upper limit of the reference range at screening or baseline), direct bilirubin > ULN (congenital nonhemolytic hyperbilirubinemia [e.g., suspicion of Gilbert's syndrome based on total and direct bilirubin] is not acceptable), creatine kinase (CK) > ULN (one repeat test allowed), thyroid stimulating hormone (TSH) outside normal range (0.75 to 5.6 mIU/L) , serum potassium outside normal range (3.5 to 5.3 mmol/L).
14. Rest sitting vital sign results abnormal and clinically significant at screening or baseline, ear temperature outside normal range, diastolic blood pressure ≥ 90 mmHg or systolic blood pressure ≥ 140 mmHg, heart rate (HR) < 55 beats/min or > 100 beats/min (test can be repeated once according to investigator's judgment).
15. Oxygen saturation (SpO2) below 95% at baseline.
16. Abnormal 12-lead ECG at screening or baseline (any test abnormality), including any of the following:

    1. QTcF > 450 ms
    2. QRS > 110 ms
    3. PR > 200 ms
    4. Second or third-degree AV block
    5. Any rhythm other than sinus rhythm of clinical significance.
17. Estimated Glomerular Filtration Rate (eGFR) < 90 mL/min (estimated using MDRD equation).
18. Participation in another clinical study of an investigational drug (or medical device) within 3 months (or 5 half-lives, whichever is longer) prior to dosing, or previous participation in any other clinical trial related to HSK3486.
19. Donation of blood within 3 months prior to screening, plasma within 2 weeks prior to screening, platelets within 6 weeks prior to screening, or receive blood products within 2 months prior to admission to the investigational site.
20. Sperm and egg donation program from screening period to 90 days after study end.
21. Pregnant or lactating women or those with positive pregnancy test results. Male or female subjects of childbearing potential did not agree to use an effective method of contraception from the time of signing ICF until 90 days after leaving the investigational site after the last dose (see Appendix 6 for details of specific contraceptive methods).
22. Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, within 30 days prior to dosing or during the clinical trial.
23. Use or intend to use of any prescription, nonprescription, vitamin, herbal, or nutraceutical within 14 days prior to dosing or during the clinical trial.
24. Smoking (≥ 5 cigarettes per day) within 6 months prior to screening, or inability to quit smoking during the trial.
25. Positive alcohol breath test, or regular drinking within 6 months prior to dosing or during the trial, i.e. drinking more than 21 units (men) or 14 units (women) of alcohol per week (1 unit =360 mL beer or 45 mL spirits or 150 mL wine at 40% alcohol).
26. Positive urine drug abuse screening (morphine, tetrahydrocannabinol, methamphetamine, methylenedioxyamphetamine, ketamine), or history of drug abuse, drug dependence within 6 months prior to screening, or drug use within 3 months prior to screening.
27. Subjects who tested positive for COVID-19 during screening.
28. Eating fruits or foods affecting metabolic enzymes, such as grapefruit (citrus), pomelo, etc., within 7 days prior to screening; and not abstaining from the above beverages, fruits or foods during the study period.
29. Previous chronic excessive consumption (more than 8 cups per day, 1 cup =250 mL) of tea, coffee or caffeinated beverages, or intake of caffeine and/or purine-rich foods or beverages (e.g. coffee, tea, chocolate, caffeinated carbonated beverages, cola, etc.) within 48 hours prior to screening, or refusal to stop drinking tea, coffee and/or caffeinated beverages during the trial.
30. Performing or unwilling to refrain from strenuous physical activity, which could cause muscle aches or injury, including contact sports, at any time from 3 days prior to dosing through the end-of- study visit.
31. Subjects who were compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical disease (e.g., infectious disease).
32. Any condition or situation that, in the opinion of the investigator, would prevent proper evaluation of the safety or efficacy of the study drug according to the study protocol (e.g., poorly compliant subject, poorly vascular condition, allergies to medical plastics/latex).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2024-04-09 (Actual); Primary Completion 2024-05-19 (Actual); Study Completion 2024-11-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Gobroad Boren Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 175 subjects were screened in this study, 112 subjects failed screening, 3 subjects did not complete all procedures or assessments for inclusion and exclusion criteria, 48 subjects were randomized, and all 48 subjects completed the study.
Groups:
- Sequence 1: C-B-A: C: HSK3486 0.4 mg/kg (Study drug) B: Moxifloxacin hydrochloride tablet 0.4g (Positive control) A: Placebo (HSK3486 simulator) (Negative control)
- Sequence 2: A-B-C: A: Placebo (HSK3486 simulator) (Negative control) B: Moxifloxacin hydrochloride tablet 0.4g (Positive control) C: HSK3486 0.4 mg/kg (Study drug)
- Sequence 3: B-C-A: B: Moxifloxacin hydrochloride tablet 0.4g (Positive control) C: HSK3486 0.4 mg/kg (Study drug) A: Placebo (HSK3486 simulator) (Negative control)
- Sequence 4: C-A-B: C: HSK3486 0.4 mg/kg (Study drug) A: Placebo (HSK3486 simulator) (Negative control) B: Moxifloxacin hydrochloride tablet 0.4g (Positive control)
- Sequence 5: A-C-B: A: Placebo (HSK3486 simulator) (Negative control) C: HSK3486 0.4 mg/kg (Study drug) B: Moxifloxacin hydrochloride tablet 0.4g (Positive control)
- Sequence 6: B-A-C: B: Moxifloxacin hydrochloride tablet 0.4g (Positive control) A: Placebo (HSK3486 simulator) (Negative control) C: HSK3486 0.4 mg/kg (Study drug)
Period: Overall Study
Arm/Group | Sequence 1: C-B-A | Sequence 2: A-B-C | Sequence 3: B-C-A | Sequence 4: C-A-B | Sequence 5: A-C-B | Sequence 6: B-A-C
Started | 8 | 8 | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1: C-B-A | Sequence 2: A-B-C | Sequence 3: B-C-A | Sequence 4: C-A-B | Sequence 5: A-C-B | Sequence 6: B-A-C | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age calculation used the date of consent form signed minus of the date of birth
  Years
    Age (Years) | 34.3 (4.77) | 31.1 (4.94) | 30.9 (3.56) | 31.0 (5.76) | 31.6 (5.26) | 34.9 (5.00) | 32.3 (4.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 1 | 0 | 2 | 8
  Male | 6 | 6 | 7 | 7 | 8 | 6 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 8 | 8 | 8 | 8 | 8 | 8 | 48
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Baseline BMI [Mean (Standard Deviation); unit: kg/m2] — Baseline BMI was defined as weight divided by height on Day1 of the first period
  kg/m2 | 22.74 (0.964) | 22.81 (2.017) | 22.88 (1.429) | 21.41 (0.777) | 23.58 (1.296) | 22.70 (1.9777) | 22.69 (1.546)

OUTCOME MEASURES:

1. Primary Outcome: Change-from-baseline in QTc Interval
Description: Corrected for HR using the individual QT correction method (QTcI) - ΔQTcI
Time Frame: From the base line ECG (D-2) to end of the period, up to 24 hours post-dose
Measure: Least Squares Mean (90% Confidence Interval); unit: ms
Groups:
- C (Study Drug): HSK3486 0.4 mg/kg (Study drug)
- B (Positive Control): Moxifloxacin hydrochloride tablet 0.4g (Positive control)
- A (Placebo): (HSK3486 simulator) (Negative control)
Arm/Group | C (Study Drug) | B (Positive Control) | A (Placebo)
Number analyzed (Participants) | 48 | 48 | 48
ms
  30s post-dose | 2.1 [0.46 to 3.74] | 5.1 [2.96 to 7.29] | -0.1 [-1.70 to 1.41]
  1 min post-dose | 4.1 [2.07 to 6.12] | -4.4 [-6.46 to -2.42] | 0.0 [-1.89 to 1.96]
  2 min post-dose | -3.1 [-4.24 to -1.90] | -7.7 [-8.88 to -6.56] | -3.1 [-4.24 to -1.91]
  3 min post-dose | -0.1 [-1.24 to 0.97] | -4.4 [-5.51 to -3.33] | -0.9 [-2.02 to 0.15]
  5 min post-dose | 4.4 [3.33 to 5.46] | -3.0 [-4.05 to -1.93] | 0.4 [-0.70 to 1.41]
  8 min post-dose | 5.1 [3.97 to 6.23] | -1.3 [-2.42 to -0.19] | 1.0 [-0.13 to 2.11]
  10 min post-dose | 4.7 [3.51 to 5.82] | -2.9 [-4.06 to -1.78] | 0.8 [-0.30 to 1.99]
  15 min post-dose | 3.3 [2.33 to 4.26] | -3.7 [-4.63 to -2.72] | 0.6 [-0.33 to 1.59]
  30 min post-dose | 1.0 [0.16 to 1.82] | -1.6 [-2.40 to -0.76] | 0.4 [-0.38 to 1.25]
  1 h post-dose | -0.1 [-1.22 to 1.12] | 5.2 [4.06 to 6.38] | 0.5 [-0.62 to 1.70]
  2 h post-dose | 1.1 [-0.07 to 2.34] | 10.0 [8.80 to 11.20] | 1.3 [0.08 to 2.46]
  3h post-dose | 0.5 [-0.75 to 1.77] | 13.2 [11.99 to 14.50] | 0.9 [-0.38 to 2.11]
  4h post-dose | 2.6 [1.30 to 3.84] | 14.8 [13.55 to 16.09] | 3.0 [1.75 to 4.27]
  6h post-dose | -1.0 [-2.98 to 0.93] | 8.0 [6.10 to 9.97] | -0.9 [-2.86 to 1.03]
  8h post-dose | -1.7 [-3.58 to 0.17] | 7.4 [5.58 to 9.29] | 1.12 [-2.41 to 1.30]
  12h post-dose | -0.9 [-2.70 to 0.91] | 6.2 [4.36 to 7.95] | 0.8 [-1.03 to 2.55]
  24h post-dose | -0.7 [-2.18 to 0.72] | 7.3 [5.85 to 8.74] | 0.1 [-1.35 to 1.52]
Statistical Analysis 1: Comparison: C (Study Drug) vs A (Placebo); 1 min post-dose; worse case for the study drug; Test type: Non-Inferiority — Upper boundary of 90% CI should not exceed the margin of 10ms; p < 0.05, Mixed Models Analysis; Mean Difference (Final Values) = 4.10, 90% CI 2-sided [1.29 to 6.82] — Upper boundary is 6.82ms, does not cross margin of the 10ms
Statistical Analysis 2: Comparison: B (Positive Control) vs A (Placebo); 3 h post-dose; worse case of the positive control; Test type: Non-Inferiority — Upper boundary of 90% CI should not exceed the margin of 10ms; p < 0.05, Mixed Models Analysis; Mean Difference (Final Values) = 12.4, 90% CI 2-sided [10.66 to 14.10] — Upper boundary is 14.10ms, cross margin of the 10ms
Statistical Analysis 3: Comparison: B (Positive Control) vs A (Placebo); 4 h post-dose, second worse case of the positive control; Test type: Non-Inferiority — Upper boundary of 90% CI should not exceed the margin of 10ms; p < 0.05, Mixed Models Analysis; Mean Difference (Final Values) = 11.8, 90% CI 2-sided [10.07 to 13.55] — Upper boundary is 13.55ms, cross margin of the 10ms

ADVERSE EVENTS:
Time Frame: From Screen period ( day -21) to 7±1 day after the last dose
Arm/Group | HSK3486( Study Drug) | Placebo | Moxifloxacin Hydrochloride
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/48 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 3/48 | 0/48 | 3/48
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HSK3486( Study Drug) (N=48) | Placebo (N=48) | Moxifloxacin Hydrochloride (N=48)
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 2 | 0 | 1
White blood cell counts decreased (Investigations) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-03-15): https://cdn.clinicaltrials.gov/large-docs/04/NCT06795204/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-11): https://cdn.clinicaltrials.gov/large-docs/04/NCT06795204/SAP_001.pdf